CLINICAL TRIAL: NCT07206225
Title: A PHASE 1, OPEN-LABEL, DOSE ESCALATION AND DOSE EXPANSION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND ANTITUMOR ACTIVITY OF PF-08052667 AS A SINGLE AGENT AND IN COMBINATION THERAPY IN PARTICIPANTS 18 YEARS OF AGE AND OLDER WITH BLADDER CANCER
Brief Title: A Study to Learn About the Study Medicine PF-08052667 in People With Bladder Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C6001001
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: NMIBC; Non-Muscle Invasive Bladder Cancer; Bladder Cancer; Bladder Tumors; Bladder Neoplasms; Malignant Tumor of Urinary Bladder; Urinary Bladder Cancer; Cancer of Bladder
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Monotherapy Dose Escalation (Experimental): PF-08052667 will be administered through intravesical instillation at defined dose levels.
  Dosing schedule is on Day 1, 8 and 15 of a 21-day cycle.
  Interventions: Drug: PF-08052667; Drug: PF-02921367
- Combination Therapy Dose Escalation (Experimental): PF-08052667 + BCG and/or sasanlimab of a 21-day cycle starting from Day 1
  Interventions: Drug: PF-08052667; Drug: Sasanlimab; Drug: BCG; Drug: PF-02921367
- Dose Optimization and Expansion (Experimental): PF-08052667 monotherapy or in combination with BCG and/or sasanlimab at dose levels/schedules for PF-08052667 determined in Parts 1 and 2.
  Interventions: Drug: PF-08052667; Drug: Sasanlimab; Drug: BCG; Drug: PF-02921367

INTERVENTIONS:
Drug: PF-08052667 — PF-08052667 will be administered intravesical (IVe) instillation following a PF-02921367 (DDM) bladder pre-wash
  Other Names: SGN-B6N
Drug: Sasanlimab — Sasanlimab will be administered as subcutaneous (SC) injection
  Other Names: PF-06801591
  Arms: Combination Therapy Dose Escalation; Dose Optimization and Expansion
Drug: BCG — BCG will be administered intravesical (IVe) instillation
  Arms: Combination Therapy Dose Escalation; Dose Optimization and Expansion
Drug: PF-02921367 — PF-02921367 (DDM) is a 10-min pre- wash and will be administered intravesical (IVe) instillation
  Other Names: DDM

SUMMARY:
The purpose of this study is to learn how a new medicine called PF-08052667 works when used by itself or together with another medicine called Bacillus Calmette Guerin (BCG), and/or a medicine called sasanlimab.

This study is for adults who have a type of bladder cancer that hasn't spread into the muscle layer of the bladder but is more likely to come back or grow. It includes people whose cancer has come back or hasn't gone away after receiving standard treatments like BCG. It may also include people who, based on their doctor's opinion, cannot receive standard treatments or those treatments are not available to them.

The study has three parts:

* Part 1 (monotherapy dose escalation) will test PF-08052667 as a single-agent at increasing dose levels in participants with certain bladder cancer whose disease has worsened on or after standard treatments.
* Part 2 (combination dose escalation) will test PF-08052667 in combination with BCG and/or sasanlimab (fixed dose) in participants with certain bladder cancer whose disease has worsened on or after standard treatments.
* Part 3 (dose optimization and expansion) will further test PF-08052667 as a single agent or in combination with BCG and/or sasanlimab, at the dose(s) based on findings from Part 1 and Part 2 in participants with certain bladder cancer including those who has never received standard treatments.

All participants will receive the study drug PF-08052667. Only participants in Part 2 and Part 3 of the study will also receive BCG and/or sasanlimab. PF-08052667 will be given as an intravesical infusion, which means it will be injected directly into the bladder. Sasanlimab will be given as a subcutaneous injection, which means it will be injected under the skin.

For all parts, treatment with study medicines will continue until either a participant has decided to stop taking part in the study or is asked to leave the study for various reasons or up to about 2 years, whichever occurs first. Duration of trial participation for each participant will vary as long-term follow-up will continue after treatment discontinuation until loss to-follow-up or death, or until the study is stopped by the sponsor.

ELIGIBILITY:
INCLUSION CRITERIA:

1. 18 years of age or older (or the minimum age of consent per local regulations)
2. Histological diagnosis of high-risk, non-muscle invasive urothelial carcinoma of the bladder defined according to the WHO grading system as carcinoma in situ (CIS), with or without concurrent T1/Ta papillary disease. Note: High-grade T1/Ta papillary disease, in the absence of CIS, may be eligible for certain cohorts in Part 2 and 3
3. BCG unresponsive and BCG-exposed cohorts should have persistent or recurrent disease after receiving at least 5 out of 6 doses of the BCG induction therapy.
4. Have refused or are ineligible or not appropriate for radical cystectomy
5. Tissue Requirement: Available tumor tissue within the last 6 months. On-treatment tumor biopsy is optional, unless mandated based on emerging data, or participating in the Biomarker Cohort, or for disease assessment
6. ECOG PS 0 or 1

EXCLUSION CRITERIA:

1. Concomitant anti-cancer therapy for Non-Muscle Invasive Bladder Cancer (NMIBC); and prior radiation therapy to the bladder are not allowed
2. Renal or hepatic impairment; and hematologic abnormalities as defined in the protocol
3. Participants with active, uncontrolled infection as specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2030-01-29 (Estimated); Study Completion 2033-01-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) in dose escalation in Part 1 and Part 2 participants only | Day of first dose (Day 1) Up to 21 days
  Any AE occurring during the DLT observation period that is attributed to PF-08052667 and not to the underlying disease or other causes is considered a DLT. DLT rate estimated based on data from DLT-evaluable participants during the DLT evaluation period.
Number of participants with adverse events (AEs) in Part 1 and Part 2 participants only | From the first day through 30-37 days after the last study treatment, up to approximately 2 years
  AEs as characterized by type, frequency, severity (CTCAE v5.0), seriousness, and relatedness to study drug(s).
Number of participants with laboratory abnormalities in Part 1 and Part 2 participants only | From the first day through 30-37 days after the last study treatment, up to approximately 2 years
  Laboratory abnormalities as characterized by type, frequency, severity
Recurrence-free survival (RFS) in Part 3 participants only | Through end of study and up to approximately 2 years
  RFS is defined as the time from the first dose until recurrence of high-grade disease, or death due to any cause, whichever occurs first
Event-free survival (EFS) in Part 3 participants only | Through end of study and up to approximately 2 years
  EFS is defined as the time from the first dose until the first occurrence of an EFS event including progressive disease, recurrence of high-grade disease, or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
PK: Maximum Observed Serum Concentration (Cmax) | From the first day through 30-37 days after the last study treatment
  Cmax of PF-08052667as a monotherapy (Part 1) and in combination with BCG and/or sasanlimab (Part 2 and Part 3)
PK: Time to Reach Maximum Observed Serum Concentration (Tmax) | From the first day through 30-37 days after the last study treatment
  Tmax of PF-08052667as a monotherapy (Part 1) and in combination with BCG and/or sasanlimab (Part 2 and Part 3)
PK: Minimum observed serum concentration (Ctrough) | From the first day through 30-37 days after the last study treatment
  Ctrough of PF-08052667as a monotherapy (Part 1) and in combination with BCG and/or sasanlimab (Part 2 and Part 3)
PK: Area under the concentration-time curve (AUC) from time zero to last (AUC from time 0 to AUClast) | From the first day through 30-37 days after the last study treatment
  AUClast of PF-08052667as a monotherapy (Part 1) and in combination with BCG and/or sasanlimab (Part 2 and Part 3)
PK: Half-life (t1/2) | From the first day through 30-37 days after the last study treatment
Incidence of Anti-Drug Antibody (ADA): Immunogenicity of PF-08052667 as a single agent (Part 1) and in combination with BCG and/or sasanlimab (Part 2 and Part 3) | Through 30-37 days after the last study treatment, up to approximately 2 years
  Incidence and titers of ADA and neutralizing antibody against PF-08052667
Duration of Complete Response (CR) in Part 1 and Part 2 participants only | Through end of study and up to approximately 2 years
  Duration of CR is the time from first documentation of CR until the first occurrence of an Event-free survival (EFS) event
Complete Response Rate (CRR) in Part 1 and Part 2 participants only | Through end of study and up to approximately 2 years
  CR rate is defined as the proportion of subjects achieving CR
Overall survival (OS) in Part 3 participants only | Through end of study approximately 5 years from last participant enrollment
  Overall survival (OS) is defined as the time from the date of first dose to the date of death due to any cause
Cystectomy-free survival in all Parts | Through end of study and up to approximately 2 years
  Cystectomy-free survival is defined as the time from the first dose until cystectomy or death due to any cause, whichever occurs first
Event-free survival (EFS) in Part 1 and Part 2 participants only | Through end of study and up to approximately 2 years
  EFS is defined as the time from the first dose until the first occurrence of an EFS event including progressive disease, recurrence of high-grade disease, or death due to any cause, whichever occurs first
Recurrence-free survival (RFS) in Part 1 and Part 2 participants only | Through end of study and up to approximately 2 years
  RFS is defined as the time from the first dose until recurrence of high-grade disease, or death due to any cause, whichever occurs first
Rate of cystectomy in all parts | Through end of study and up to approximately 2 years
  Rate of cystectomy is defined as the proportion of participants who had a cystectomy while on study
Number of participants with adverse events (AEs) in Part 3 participants only | From the first day through 30-37 days after the last study treatment, up to approximately 2 years
  AEs as characterized by type, frequency, severity (CTCAE v5.0), seriousness, and relatedness to study drug(s)
Number of participants with laboratory abnormalities in Part3 participants only | From the first day through 30-37 days after the last study treatment, up to approximately 2 years
  Laboratory abnormalities as characterized by type, frequency, severity

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (27):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Hematology/Oncology - Westwood (Building 300), Los Angeles, California
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas - Clinical Research Center, Fairway, Kansas
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Upstate Specialty Services at Harrison Center, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical University-Community Campus, Syracuse, New York
  - Duke Cancer Institute, Durham, North Carolina
  - AUC Urologists, LLC, Myrtle Beach, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Grand Strand Medical Center, Myrtle Beach, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - Coastal Eye Group, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - UT Southwestern Medical Center-William P. Clements Imaging Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baptist M&S Imaging (Medical Center), San Antonio, Texas
  - USA Clinical Trials, San Antonio, Texas
  - MCOA Eye Associates, San Antonio, Texas
- France (2):
  - Pitie Salpetriere University Hospital, Paris, Other
  - Gustave Roussy, Villejuif, Other
- Israel (4):
  - Rambam Health Care Campus, Haifa, Other
  - Hadassah Medical Center, Jerusalem, Other
  - Rabin Medical Center, Petah Tikva, Other
  - Sheba Medical Center, Ramat Gan, Other
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul, Other
  - Samsung Medical Center, Seoul, Other
- Spain (2):
  - Fundació Puigvert, Barcelona, Other
  - Hospital Universitario 12 de Octubre, Madrid, Other
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, Other, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6001001